CLINICAL TRIAL: NCT06714708
Title: SPARK: Safety and Efficacy of Low Dose Radiotherapy Combined With Sintilimab and Platinum Based Chemotherapy as Neoadjuvant Therapy for Stage II-III Non-Small Cell Lung Cancer
Brief Title: Low Dose Radiotherapy Combined With Sintilimab and Chemotherapy as Neoadjuvant Therapy for Stage II-III NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shuanghu Yuan, Professor, Anhui Provincial Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARK; CRTOG2401 (Other: CRTOG)
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: NSCLC; Neoadjuvant Immunotherapy; Low Dose Radiotherapy; Sintilimab
Keywords: NSCLC; Neoadjuvant Immunotherapy; Low Dose Radiotherapy; Sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Radiotherapy combined with Sintilimab and Chemotherapy (Experimental): Neoadjuvant treatment：two cycles of sintilimab and platinum based chemotherapy，simultaneously undergoing radiotherapy 30Gy/15F
  Interventions: Radiation: Experimental
- Sintilimab in combination with Chemotherapy (Active Comparator): Neoadjuvant treatment：two cycles of sintilimab and platinum based chemotherapy
  Interventions: Drug: Active comparator

INTERVENTIONS:
Radiation: Experimental — Radiation: 30Gy/15F Drug: Sintilimab, 200mg IV D1 Q3W Drug: Cisplatin, 75mg/m2 D1 IV Q3W or Carboplatin AUC 5-6mg/ml/min D1 IV Q3W Drug: Pemetrexed, 500mg/m2 D1 IV Q3W or Albumin paclitaxel 260mg/m2，D1 or 130mg/m2，D1,8 IV Q3W
  Arms: Low Dose Radiotherapy combined with Sintilimab and Chemotherapy
Drug: Active comparator — Drug: Sintilimab, 200mg IV D1 Q3W Drug: Cisplatin, 75mg/m2 D1 IV Q3W or Carboplatin AUC 5-6mg/ml/min D1 IV Q3W Drug: Pemetrexed, 500mg/m2 D1 IV Q3W or Albumin paclitaxel 260mg/m2，D1 or 130mg/m2，D1,8 IV Q3W
  Arms: Sintilimab in combination with Chemotherapy

SUMMARY:
To evaluate efficacy and safety of low dose radiotherapy combined with sintilimab and platinum based chemotherapy as neoadjuvant therapy for stage II-III Non-Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following inclusion criteria are eligible for inclusion in this study:

  1. Sign a written Informed Consent Form (ICF) and be able to comply with the visit and related procedures specified in the protocol.
  2. Age ≥ 18 years old.
  3. Primary non-small cell lung cancer (including adenocarcinoma and squamous cell carcinoma) diagnosed by cytology or histology.
  4. According to the International Association for the Study of Lung Cancer and the Joint Committee on Cancer Classification 8th edition (AJCC8) TNM staging classification of lung cancer, the clinical staging is IIB (primary tumor>4cm), IIIA, or IIIB (resectable N2 only) stage. Resectable N2 refers to non bulk (defined as a short diameter less than 3cm), discrete, or single site N2 involvement. If clinically suspected as N2 or N3, pathological confirmation is required.
  5. Non squamous NSCLC subjects need to undergo genetic testing to confirm the absence of EGFR sensitive mutations and ALK rearrangements. Squamous NSCLC subjects are not required to undergo genetic testing, but subjects with known EGFR sensitive mutations and ALK rearrangements should not be included in the study.
  6. Considered suitable for radical resection surgery.
  7. The lung function meets the criteria for planned lung resection (FEV1 ≥ 50% predicted value, MVV ≥ 50% predicted value), and there are no surgical contraindications.
  8. Can provide sufficient tissue specimens that meet the requirements for PD-L1 testing during the screening period.

According to RECIST V1.1, there is at least one measurable lesion. 10. The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score is 0 or 1.

11. Have not received any systemic anti-tumor therapy or local radiotherapy for NSCLC in the past.

12. Possess sufficient organ and bone marrow function, with laboratory test values meeting the following requirements within 7 days prior to enrollment (no blood components, cell growth factors, albumin, or other intravenous or subcutaneous drugs for correcting hematological or liver and kidney dysfunction are allowed within 14 days prior to obtaining laboratory tests), as follows: Hematological function is sufficient, defined as absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, hemoglobin ≥ 100g/L;

* Adequate liver function, defined as total bilirubin levels ≤ 1.5 × upper limit of normal (ULN) and levels of aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN, albumin (ALB) ≥ 35g/L;
* Adequate renal function, serum creatinine (Scr) ≤ 1.5 × ULN, creatinine clearance rate (CrCl) ≥ 60mL/min (calculated using the Cockcroft/Gault formula), and urine routine test results showing urinary protein (UPRO)<2+or 24-hour urine protein dose<1g; Within 7 days prior to treatment, the international normalized ratio (INR) is ≤ 1.5 × ULN, and the prothrombin time (PT) or activated partial thromboplastin time (APTT) is ≤ 1.5 × ULN.

  13. For female subjects of childbearing age, urine or serum pregnancy tests were negative within 7 days prior to receiving the first study drug administration. 14.If the urine pregnancy test result is positive, a blood pregnancy test is required.

  15.If there is a risk of conception, male and female patients should use highly effective contraception (i.e. methods with an annual failure rate of less than 1%) and continue for at least 180 days after stopping the trial treatment. Note: If abstinence is the subject's usual lifestyle and preferred contraceptive method, then abstinence is acceptable as a contraceptive method.

Exclusion Criteria:

* 1. Histological and pathological examinations show the presence of coexisting small cell carcinoma, large cell neuroendocrine tumor, and sarcomatoid tumor components.

  2. Tumors invade the diaphragm, mediastinum, heart, pericardium, large blood vessels (such as aorta), trachea, recurrent laryngeal nerve, esophagus, vertebral body, and protuberance.

  3. Tumor of the superior sulcus of the lung. 4. There are tumor nodules in the contralateral lung lobe; If there is clinical suspicion of tumor nodules in the contralateral lung lobe, biopsy is required for clarification.

  5. Confirm or suspect patients with brain metastases. 6. Currently participating in interventional clinical research treatment, or having received other investigational drugs or devices within the first 4 weeks of randomization.

  7. Previous use of anti-PD-1, anti-PD-L1, anti programmed death receptor ligand 2 (PD-L2), or anti cytotoxic T lymphocyte associated antigen 4 (CTLA-4) drugs or any other drugs that act on T cell co stimulatory or immune checkpoint pathways (such as OX40, CD137, etc.) and adoptive cell immunotherapy.

  8. Have received Chinese herbal medicine, traditional Chinese patent medicines and simple preparations with anti-tumor indications, or drugs with immunomodulatory effects (including thymic peptides, interferon, interleukin) within the first two weeks of randomization.

  9. Have undergone major surgery within the first 4 weeks of randomization. 10. There are unhealed surgical incisions, ulcers, or fractures present. 11. Received attenuated live vaccine within the first 4 weeks of randomization (or planned to receive attenuated live vaccine during the study period). Note: Accepting inactivated virus vaccines for injection against seasonal influenza is allowed; However, receiving attenuated live influenza vaccines is not allowed.

  12. Patients who require long-term systemic use of corticosteroids; Received any other form of immunosuppressive therapy within the first 7 days of randomization. Note: Local corticosteroids administered via nasal spray, inhalation, or other routes, or systemic corticosteroids at physiological doses (≤ 10mg/day of prednisone or equivalent), or for pre-treatment purposes (such as preventing contrast agent allergies), are allowed.

  13. There is a history of non infectious pneumonia requiring glucocorticoid treatment or current interstitial lung disease within the previous year of randomization.

  14. Within the first 2 years of randomization, there have been active autoimmune diseases that require systemic treatment (such as the use of disease improving drugs, corticosteroids, or immunosuppressants), including but not limited to inflammatory bowel disease, such as ulcerative colitis or Crohn's disease; Diverticulitis; Celiac disease; Systemic lupus erythematosus; Sarcoidosis syndrome or Wegener syndrome (granulomas with polyangitis); Graves' disease; Rheumatoid arthritis; Multiple sclerosis; Vasculitis; Glomerulonephritis; Antiphospholipid syndrome; Pituitary inflammation; Uveitis, etc. Alternative therapies such as thyroid hormone, insulin, or physiological dose corticosteroids used for adrenal or pituitary insufficiency are not considered systemic treatments. Patients with positive autoimmune antibodies need to be evaluated and confirmed by the researcher that there are no autoimmune diseases that require systemic treatment before they can be enrolled.

  15. Suffering from primary immunodeficiency disease. 16. Past or current presence of myocarditis. 17. Prior to randomization, there was insufficient recovery from toxicity and/or complications caused by any intervention measures (i.e.,>grade 1 or not recovered to baseline levels).

  18. ≥ Grade 2 peripheral neuropathy. 19. Genetic bleeding tendency or coagulation dysfunction, or history of thrombosis: Any arterial thrombosis, embolism, or ischemia occurred within the first 6 months of randomization, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism. A history of deep vein thrombosis or any other severe thromboembolism within the first 3 months of randomization (implantable venous infusion port or catheter-related thrombosis, or superficial vein thrombosis is not considered a "severe" thromboembolism).

  20. Uncontrolled hypertension (systolic blood pressure greater than 160mmHg and/or diastolic blood pressure greater than 100mmHg); History of hypertensive crisis or hypertensive encephalopathy; Uncontrolled hyperglycemia (fasting blood glucose>8.9 mmol/L).

  21. Any unstable systemic disease or concurrent disease, including but not limited to:
  * Active infection (requiring treatment with anti infective drugs or having used systemic anti infective drugs within the week prior to randomization);
  * Congestive heart failure [New York Heart Association (NYHA) classification ≥ II]; Serious arrhythmias, liver, kidney or metabolic diseases that require medication treatment;
  * Untreated coronary atherosclerotic heart disease; Type I or II respiratory failure; History of gastrointestinal perforation and/or fistula, intestinal obstruction, extensive intestinal resection, or long-term chronic diarrhea within the past 6 months.

    22. Received solid organ or blood system transplantation. 23. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV1/2 antibody positive), known active syphilis.

    24. Active or tuberculosis requiring medical intervention at this stage, including but not limited to tuberculosis.

    25. Active hepatitis B.
  * Subjects with hepatitis B who meet the following criteria meet the inclusion criteria: HBsAg (+) or HBcAb (+), HBV viral load before randomization<1000 copies/ml or<200IU/ml or lower than the detection limit.

HBsAg (+) subjects should receive anti HBV therapy throughout the entire study drug treatment period to avoid viral activation.

For subjects with anti HBc (+), HBsAg (-), anti HBs (-), and HBV viral load (-), prophylactic anti HBV treatment is not necessary, but close monitoring of virus reactivation is necessary.

26. Active hepatitis C (HCV antibody positive and HCV-RNA level above the detection limit).

27. Malignant tumors other than diagnosed NSCLC within the first 5 years of randomization, excluding fully treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, and papillary thyroid carcinoma after radical surgery.

28. It is known that there is an allergic reaction to the active ingredients and/or any excipients of the selected chemotherapy regimen (non squamous NSCLC: pemetrexed plus cisplatin or carboplatin; squamous NSCLC: gemcitabine, docetaxel, paclitaxel or albumin paclitaxel plus cisplatin or carboplatin).

29. Pregnant or lactating women or women preparing to become pregnant or breastfeed during the study period.

30. It is known that there are mental illnesses or drug abuse situations that may affect compliance with experimental requirements, and there is a history of alcohol abuse.

31. There may be medical history, diseases, treatments, or laboratory abnormalities that could interfere with the trial results, hinder the full participation of the subjects in the study, or the researcher believes that participating in the study is not in the best interests of the subjects. Local or systemic diseases caused by non malignant tumors, or secondary reactions to cancer, can lead to higher medical risks and/or uncertainty in survival evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response（pCR） rate | up to 8 weeks after surgery
  Pathological complete response (pCR) rate is defined as the proportion of participants whose tumor in the stomach and lymph node completely disappeared, as determined by a pathologist.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | up to 8 weeks after surgery
  Major pathological response (MPR) rate is defined as the proportion of participants whose percentage of residual tumor in the stomach and lymph node decreased to < 10%, as determined by a pathologist.
Objective Response Rate （ORR） | through study completion, an average of 1 year
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
Event Free Survival（EFS） | up to 3 years
  proportion of participants who have no events，including death, disease progression, change of chemotherapy regimen, switching to chemotherapy, addition of other treatments, occurrence of lethal or intolerable side effects, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Cancer Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Background] Li J, Lu S, Tian Y, Jiang L, Li L, Xie SH, Li Q. Neoadjuvant low-dose radiotherapy plus durvalumab and chemotherapy for potentially resectable stage III NSCLC: A phase Ib dose-escalation study. Radiother Oncol. 2024 Jul;196:110316. doi: 10.1016/j.radonc.2024.110316. Epub 2024 Apr 26. PMID 38679201